CLINICAL TRIAL: NCT06487949
Title: Comparative Analysis of Valsartan 80 mg and Amlodipine 5 mg in Fixed-Dose Combination Therapy Versus Combination Free Drug Therapy for Ambulatory Blood Pressure Management: A Randomized Controlled Trial
Brief Title: Valsartan and Amlodipine in Blood Pressure Management: Fixed-Dose vs. Free Drug Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1400.505
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
Keywords: hypertension; 24 hours ambulatory blood pressure monitoring; fix dose combination
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- valsartan- Amlodipine fix dose combination pill (Experimental): Patients with hypertension eligible receiving valsartan- Amlodipine 80/5 mg fix dose combination (FDC) pill
  Interventions: Drug: valsartan-amlodipine 80/5 mg FDC
- Valsartan- Amlodipine free dose combination (Active Comparator): Patients with hypertension eligible receiving valsartan 80 mg and amlodipine 5 mg as free dose of drugs separately
  Interventions: Drug: valsartan 80 mg and amlodipine 5 mg as free combination

INTERVENTIONS:
Drug: valsartan-amlodipine 80/5 mg FDC — fix dose combination of valsartan 80 mg and Amlodipine 5 mg given as single pill
  Other Names: FDC
  Arms: valsartan- Amlodipine fix dose combination pill
Drug: valsartan 80 mg and amlodipine 5 mg as free combination — Free combination of valsartan 80 mg and amlodipine 5 mg given separately
  Other Names: free drug combination
  Arms: Valsartan- Amlodipine free dose combination

SUMMARY:
Patients aged 35 to 70 years with newly diagnosed stage 1 or 2 hypertension ( HTN) was randomized to receive either Valsartan 80 mg/Amlodipine 5 mg fix dose combination (FDC) or a free equivalent combination. Ambulatory blood pressure monitoring at baseline and 8 weeks post-treatment initiation was performed.

DETAILED DESCRIPTION:
Patients were eligible for enrollment if they were between 35 and 70 years old and diagnosed with stage 1 or 2 hypertension at the time of enrollment, according to the 2017 ACC/AHA Guidelines (systolic blood pressure > 130 mmHg and/or diastolic blood pressure > 80 mmHg), and required the initiation of antihypertensive medications.

This study used the permutation block randomization method (block size = 4) for the randomization process.Patients were randomly assigned to either the FDC group or the free equivalent combination group.

Eligible patients underwent an 8-week period during which they received either Valsartan 80 mg and Amlodipine 5 mg as an FDC or as free equivalent combinations. The FDC group received one single tablet daily, while the free combination group received the medications on separate tablets (amlodipine daily and Valsartan in the evening). 24-hour ambulatory blood pressure monitoring (ABPM) at the time of inclusion and at the end of the 8-week period were performed using a standard ABPM device that the patients wore with an appropriately sized cuff.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage 1 or 2 hypertension at the time of enrollment, according to the 2017 ACC/AHA Guidelines (systolic blood pressure > 130 mmHg and/or diastolic blood pressure > 80 mmHg), and required the initiation of antihypertensive medications

Exclusion Criteria:

* Patients previously been on antihypertensive drugs
* Patients had secondary high blood pressure
* Patients had severe high blood pressure (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg)
* Patients had ischemic heart disease in the past
* Patients were unable to receive any part of the treatment
* Patients who refuse to take part in study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Mean 24 hours systolic blood pressure | 8 weeks
  The average systolic blood pressure over 24 hours, during the day and at night
Mean 24 hours diastolic blood pressure | 8 weeks
  The average diastolic blood pressure over 24 hours, during the day and at night
Mean 24 hours mean blood pressure | 8 weeks
  The average mean blood pressure over 24 hours, during the day and at night

SECONDARY OUTCOMES:
Dipping | 8 weeks
  Drop of Mean systolic pressure more than 10% during nights compare to mean systolic pressure at days

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
The data is available based on rational request